CLINICAL TRIAL: NCT03252912
Title: Cerebrospinal Fluid Biomarkers Value: Exploratory and Prospective Study in Leptomeningeal Metastases of Breast Cancer (LCS Bio Sein)
Brief Title: Study in Leptomeningeal Metastases of Breast Cancer
Acronym: LCS Bio Sein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICM-URC 2015/71
Record Dates: First submitted 2017-08-10; First posted 2017-08-17 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological samples (Experimental): The CSF samples will be taken at the occasion of the first lumbar puncture performed for clinical purposes (suspected LM). If necessary for the routine diagnosis, a second and a third lumbar puncture will be performed according to the gold standard Two EDTA tubes (5 mL) and two dried tubes (5mL) will be will be taken the same day as the first lumbar puncture and transferred at ambient temperature to the Biological Resource Center of the ICM (Jean-Pierre Bleuse, Biobank number BB-0033-00059) to be processed within 1 hour Blood samples will be centrifuged at 3,000 g for 10 minutes at ambient temperature and will be aliquoted in 4 plasma and 4 serum aliquots and then stored at -80°C. Aliquots must be anonymized.
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples — Two EDTA tubes (5 mL) and two dried tubes (5mL) will be will be taken the same day as the first lumbar .

SUMMARY:
Breast cancer (BC) is the most frequent cause of leptomeningeal metastases (LM) .As for brain parenchymal metastases, the incidence of LM seems to be increasing, due to the growing incidence of metastatic BC, the improvement of survival and the poor diffusion of therapeutic agents into the central nervous system (CNS). Several prognostic factors have been identified, including the age at diagnosis, the functional and neurological status, the delay between the diagnosis of cancer and that of LM. The survival of patients is poor, less than 6 months in most published series. Several neuronal biomarkers could also be good candidates, such as the neurogranin CSF and/or serum levels or the CNS neurofilaments (NF), that seem to be a good reflect of axonal injury and neuronal loss. CNS NF have been investigated in several neurological diseases including Alzheimer's disease, Parkinson's disease, amyotrophic lateral sclerosis and multiple sclerosis, but not yet in CNS metastases. Indeed, the creation of a clinico-biological collection seems to be of high value in order to investigate future biomarkers of interest

DETAILED DESCRIPTION:
Breast cancer (BC) is the most frequent cause of leptomeningeal metastases (LM). As for brain parenchymal metastases, the incidence of LM seems to be increasing, due to the growing incidence of metastatic BC, the improvement of survival and the poor diffusion of therapeutic agents into the central nervous system (CNS). Several prognostic factors have been identified, including the age at diagnosis, the functional and neurological status, the delay between the diagnosis of cancer and that of LM. Other CSF biomarkers have been evaluated for the diagnosis of leptomeningeal metastases. Finally, the CellSearch® technique allows for the characterisation of proteins expressed by CSF tumors cells (E.G., HER2) and will make possible a better understanding of the physiopathology of tumor dissemination to the CS.

Other neuronal biomarkers could be interesting for the diagnosis of LM in BC patients. Among them, the protein Tau (total-Tau or T-Tau) is involved in several neurological diseases. However, to date, no study has evaluated CSF or serum T-Tau in LM from solid tumors.

Several neuronal biomarkers could also be good candidates, such as the neurogranin CSF and/or serum levels or the CNS neurofilaments (NF), that seem to be a good reflect of axonal injury and neuronal loss.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥ 18 years-old, no age limit;
2. Histologically confirmed diagnosis of BC;
3. Hormone receptors and HER2 statuses of the primary tumor available;
4. Suspected LM based on clinical symptoms or signs, or radiological abnormalities;
5. Indication of diagnosis lumbar puncture decided by the oncologist in charge of the patient;
6. Patients must be affiliated to a Social Security System;
7. Patient information and written informed consent form signed prior to any study specific procedures.

Exclusion Criteria:

1. History of other cancer(s) than the BC (except completely resected non-melanoma skin cancer or successfully treated in situ carcinoma).
2. Hormone receptors and/or HER2 statuses of the primary tumor not available;
3. Patients with a medical contra-indication to the realization of a lumbar puncture;
4. Patients with psychological, family, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule;
5. Patients who are pregnant or breast-feeding.
6. Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the CellSearch® technique on CSF samples in comparison with the conventional cytology on one to three CSF sample | through study completion, an average of 2 years
  analysis of result with the 2 technical procedure

CONTACTS AND LOCATIONS:
Overall Officials: marc ychou, Study Director — institut régional du Cancer de Montpellier
Locations (1):
- Institut régional du Cancer de Montpellier, Montpellier, France